CLINICAL TRIAL: NCT02099370
Title: A Single-center Prospective Measurement of Adherence to Treatment With Tecfidera™ in Multiple Sclerosis Patients.
Brief Title: Adherence to Treatment With Tecfidera™ in Multiple Sclerosis Patients
Acronym: ADIMS
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Derrick Scott Robertson, MD, Multiple Sclerosis Center Director, University of South Florida
Other Study IDs: US-BGT-13-10458
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Tecfidera(R); Oral medication; Adherence
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are measuring the adherence rates of an oral MS drug that is to be administered twice-daily. The investigators would like to observe any patterns that might indicate factors that greatly affect adherence.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law (e.g., Protected Health Information [PHI]).
* Aged 18 at the time of informed consent.
* Must have a relapsing form of MS.
* Male subjects and female subjects of child-bearing potential (including female subjects who are not post-menopausal for at least 1 year) must be willing to practice effective contraception (as defined by the investigator) during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Exclusion Criteria:

* Progressive form of MS
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity.
* Female subjects considering becoming pregnant while in the study.
* Female subjects who are currently pregnant or breast-feeding.
* Unwillingness or inability to comply with the requirements of the protocol including the presence of any conditional (physical, mental or social) that is likely to affect the subject's ability to comply with the protocol.
* Any other reason that, in opinion of the Investigator and/or the Sponsor, the subject is determined to be unsuitable for enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample of Multiple Sclerosis patients started on Tecfidera
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
adherence rates to Tecfidera | over one year

CONTACTS AND LOCATIONS:
Locations (1):
- USF Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida, United States